CLINICAL TRIAL: NCT00946062
Title: The Impact of Orientation and Mobility Training on Mobility, Participation and Quality of Life in Older Adults With Visual Impairments: a Randomised Controlled Trial
Brief Title: Evaluation of a Standardised Orientation and Mobility Training in Older Adults With Low Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 07-3-057.5/pl; ZonMw 94305004
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Low Vision; Aged
Keywords: low vision; ophthalmology; randomised controlled trial; mobility; orientation; cane; aged
MeSH Terms: conditions — Vision, Low; Orientation, Spatial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- regular O&M-training (Active Comparator): orientation and mobility training in use of the identification cane as provided by mobility trainers
  Interventions: Other: orientation and mobility training
- standardised O&M-training (Experimental): standardised orientation and mobility training in use of the identification cane as provided by mobility trainers who received instruction in using the standardised protocol
  Interventions: Other: orientation and mobility training

INTERVENTIONS:
Other: orientation and mobility training — orientation and mobility training

SUMMARY:
The purpose of this study is:

1. to develop a standardised orientation and mobility training (O&M-training) in the use of an identification/symbol cane by older adults with low vision, and;
2. to evaluate this newly developed standardised O&M-training with respect to effectiveness and feasibility in a randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 years or over
* Low vision
* Living independently in the community or in a home for older people
* Able to see large obstacles and to go outside for a short walk or doing groceries
* One of the following:

  1. experiencing difficulties with safely crossing a street
  2. experiencing difficulties with recognising acquaintances outdoors
  3. willing to become recognisable as being partially sighted by using the identification cane
* Written informed consent
* Orientation and Mobility training (O&M-training) in the use of an identification cane

Exclusion Criteria:

* Cognitive impairment (a score of less than 4 on the Abbreviated Mental Test 4)
* Language or hearing problems that impede completing an interview by telephone
* Confinement to bed or possible nursing home admission that impede completion of the O&M-training
* Permanent use of a walking aid incompatible with the use of an identification cane
* Having recently received an O&M-training in the use of an identification cane and permanent use of this cane

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
activities of daily life (subscale of the Groningen Activity Restriction Scale (GARS)) | 5 and 17 weeks
distance activities and mobility (subscales of the Visual Functioning Questionnaire (VFQ)) | 5 and 17 weeks

SECONDARY OUTCOMES:
activities index (Frenchay Activities Index (FAI)) | 5 and 17 weeks
social support interactions (Social Support List (SSL 12-I)) | 5 and 17 weeks
health-related quality of life (EuroQol 5D (EQ5D)) | 5 and 17 weeks
mental health and dependency (subscale of the Visual Functioning Questionnaire (VFQ)) | 5 and 17 weeks
feelings of anxiety (anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A)) | 5 and 17 weeks
symptoms of depression (depression subscale of the Hospital Anxiety and Depression Scale (HADS-D)) | 5 and 17 weeks
concerns about falling (falls efficacy scale international (FES-I)) | 5 and 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: G.I.J.M. Kempen, PhD, Principal Investigator — Maastricht University, CAPHRI School for Public Health and Primary Care
Locations (3):
- Netherlands (3):
  - Sensis, Grave
  - Royal Visio, Huizen
  - Bartimeus, Utrecht

REFERENCES:
- [Derived] Ballemans J, Zijlstra GA, van Rens GH, Schouten JS, Kempen GI. Usefulness and acceptability of a standardised orientation and mobility training for partially-sighted older adults using an identification cane. BMC Health Serv Res. 2012 Jun 8;12:141. doi: 10.1186/1472-6963-12-141. PMID 22681932
- [Derived] Zijlstra GA, van Rens GH, Scherder EJ, Brouwer DM, van der Velde J, Verstraten PF, Kempen GI. Effects and feasibility of a standardised orientation and mobility training in using an identification cane for older adults with low vision: design of a randomised controlled trial. BMC Health Serv Res. 2009 Aug 27;9:153. doi: 10.1186/1472-6963-9-153. PMID 19712448